CLINICAL TRIAL: NCT01159210
Title: An International, Multi-centre, Prospective, Open-Label, Non-Randomised, Uncontrolled Study to Assess the Efficacy and Safety of Prothromplex Total in Oral Anticoagulant Reversal in Patients With Acquired Deficiency of Prothrombin Complex Coagulation Factors (II, VII, IX, X)
Brief Title: Efficacy and Safety of Prothromplex Total (Prothrombin Complex Concentrate) in Oral Anticoagulant Reversal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 220901; 2010-019250-41 (EudraCT Number)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Prothrombin Complex Factor Deficiency
MeSH Terms: interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Prothrombin complex concentrate (coagulation factors IX, II, VII and X in combination) — Intravenous infusion; regimen is guided by the pre-treatment international normalised ratio (INR); dosage and duration of replacement therapy depend on the severity of the disorder, on the location and extent of bleeding and on the patient´s clinical condition.
  Other Names: Prothromplex Total

SUMMARY:
The purpose of the study is to assess the efficacy and safety of Prothromplex Total as a treatment for the immediate reversal of oral anticoagulant therapy with vitamin K antagonists in patients with acquired deficiency of prothrombin complex coagulation factors (II, VII, IX, X). Upon enrolment, subjects will receive Prothromplex Total for the treatment of acute bleeding due to oral anticoagulants or for the prevention of excessive bleeding during the interventional procedure (Day 1). Additional doses of Prothromplex Total may be administered at the discretion of the investigator. Efficacy and safety assessments will be performed during a period of 72 (± 4) hours after administration of the last dose of Prothromplex Total or until discharge from hospital, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 16 years or older at enrolment with acquired deficiency of prothrombin complex coagulation factors (II, VII, IX, X), due to oral anticoagulation with vitamin K antagonists (e.g. coumarin, warfarin), requiring reversal of oral anticoagulation for urgent surgery, or invasive procedure or acute bleeding episode
* Subject or parent/legally authorised representative has provided written informed consent
* Subject has INR >= 2,0 at screening
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subject has laboratory and/or clinical symptoms which are clearly indicative of overt disseminated intravascular coagulation (DIC)
* Subject has been treated with whole blood, fresh frozen plasma (FFP), or platelets within 6 hours prior to study enrolment
* Subject has a hypersensitivity to prothrombin complex concentrate (PCC) constituents (including heparin-induced thrombocytopenia)
* Subject has blood loss of >= 5 units of blood
* Subject has hereditary thrombophilia or bleeding disorder
* Subject has a life expectancy of < 3 months
* Subject has been on oral anticoagulant treatment for a period of < 4 weeks for the treatment of a thrombotic event such as deep vein thrombosis or pulmonary embolism
* Subject has an acute ischemic cardiovascular disorder
* Subject has or is suspected to have sepsis
* Subject with acute or chronic liver failure (hepatic cirrhosis Child-PUGH score C)
* Subject has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrolment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-07-09 (Actual); Primary Completion 2012-04-07 (Actual); Study Completion 2012-04-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve normalisation of International normalised ratio (INR) to <= 1.3 within 30 (±5) minutes post administration of Prothromplex Total | within 35 minutes after administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- Austria (3):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Universitätsklinik für Innere Medizin I (University Hospital for Internal Medicine I), Allgemeines Krankenhaus der Stadt Wien (General Hospital Vienna), Vienna
  - Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhügel, Vienna
- Hungary (3):
  - DEOEC, University of Debrecen, Medical and Health Science Centre, Debrecen
  - Fejer Megyei Szent György Korhaz, Székesfehérvár
  - Veszprem Megyei Csolnoky Korhaz Nonprofit Zrt., Belgyógyászati Centrum, Haematológiai Részleg, Veszprém